CLINICAL TRIAL: NCT06430853
Title: Psychobiological Effects of Lifestyle Interventions in Pregnancy
Brief Title: Psychobiological Interventions in Pregnancy
Acronym: PIP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Danielle Panelli, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-74741; 1K23HD113845 (NIH)
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Complications; Mental Health Issue; Depression, Anxiety; Pregnancy, High Risk; Biological Clock Disturbance
Keywords: Pregnancy; Stress; Mental health; Depression; Anxiety; Telomeres; Cortisol; Physical activity; Exercise
MeSH Terms: conditions — Pregnancy Complications; Depression; Anxiety Disorders; Chronobiology Disorders; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual step count (Placebo Comparator): Participants will wear an Actigraph accelerometer watch, but not be given a step count goal, between 20 and 36 weeks of gestation.
  Interventions: Device: Actigraph watch
- Step count goal (Experimental): Participants will be given a daily step count goal of 8,000 steps per day based on the Actigraph watch, between 20 and 36 weeks of gestation. If they are not at goal, a step-up protocol will be designed for each participant and reviewed with a study team member every 2 weeks.
  Interventions: Behavioral: Step count goal; Device: Actigraph watch

INTERVENTIONS:
Behavioral: Step count goal — The step count goal will be discussed at the beginning of the study, and participants will be able to see their step count on the Actigraph watch to facilitate achieving this goal. All participants will receive weekly reminders that are tailored for their intervention arm. Intervention group participants will also receive a step count diary with motivational ideas of how to obtain step goals, which will be reviewed with a study team member every 2 weeks.
  Arms: Step count goal
Device: Actigraph watch — Both groups will wear the watch. Adherence will be assessed via step counts from accelerometer watch.
  Other Names: Actigraph GT9X Link Accelerometer

SUMMARY:
This randomized control trial will evaluate whether a physical activity intervention can improve mental health and biologic markers of stress in pregnant people with depressive or anxiety symptoms. The study will enroll participants if they are presenting for prenatal care at Stanford Children's Health Obstetrics Clinic with a singleton gestation.

DETAILED DESCRIPTION:
Study Design This will be a randomized, parallel group, unblinded, single site superiority trial evaluating the impact of a physical activity intervention on reducing symptoms in people with known or screen-positivity for depression or anxiety during pregnancy. Participants will be randomized to a step count intervention versus usual care. Adherence will be monitored via Actigraph Link GT9X accelerometer watches.

Primary outcome: The primary outcome will be the mean within-person change in EPDS score between Time 2 (randomization) and Time 3 (37 weeks).

Secondary outcomes: Secondary outcomes will include additional psychobiologic measures, pregnancy complications, SMM events, and neonatal outcomes as shown below:

* Maternal Psychologic and Clinical: For psychologic measures, within person change in EPDS anxiety subscale score between Time 2 and Time 3, STAI score between Time 2 and Time 3, as well as within person change in both EPDS and STAI from Time 2 and Time 4 (6 weeks postpartum), will be assessed. Delivery outcomes (e.g. mode of delivery, gestational age at delivery) as well as complications including hypertensive disorders and SMM indicator events will be abstracted from the medical record.
* Maternal Biologic: For biologic measures, within person change in leukocyte telomere length and hair cortisol level from Time 2 and Time 3 will be assessed. Saliva samples for telomeres will be retained until the study is complete, at which point DNA will be extracted from leukocytes and telomere length will be measured using quantitative polymerase chain reaction. All correlated samples will be analyzed on the same 96-well plates. Telomere length results are reported as telomere "T" to single copy gene "S" standardized ratios which can be converted to base pairs using a standard equation. Within-person correlation of repeated continuous measures will be assessed using generalized estimated equations to evaluate longitudinal changes. Hair cortisol will be measured in two 3-inch hair sections, one at Time 2 and one at Time 3.
* Infant: Birthweight, Apgar scores, neonatal ICU admission, and length of stay will be evaluated.

Covariates: Demographic, clinical, and socioeconomic covariates of interest will be collected from participants. These variables will be ascertained via patient report (e.g. highest level of education, annual income, number of jobs worked, self-identified race and ethnicity, engagement in mental health treatments) and via chart abstraction (e.g. medical comorbidities, substance use, body mass index, neonatal birthweight and Apgar score). If covariates are unbalanced between groups, results from Aim 1 will be used to prioritize which covariates should be accounted for in adjusted models.

Analyses. The primary analysis will compare the difference in mean within person EPDS score change between Time 2 and Time 3 in the study across the control and intervention groups. If the mean EPDS differences are normally distributed, analysis will be conducted using independent t-tests. If not, analysis will be conducted using nonparametric tests such as Wilcoxon rank-sum tests. If any demographic or clinical characteristic emerges unbalanced between the randomization groups, an additional analysis will be conducted adjusting for this as a potential confounder as long as assumptions are met for linear regression techniques. Secondary outcomes will be compared using t-tests for normally distributed continuous variables, Wilcoxon rank sum tests for nonparametric continuous variables, and chi square tests for categorical variables. Changes in secondary questionnaire outcomes over time (such as differences in STAI, EPDS) will be compared using the differences in an individual's scores. Mean maternal leukocyte telomere and hair cortisol differences between Time 2 and Time 3 will be compared across groups as continuous variables.

Missing data: Based on our prior longitudinal studies with similar populations, we expect completion rates of >70%, with little item-level missing data. We will conduct intent-to-treat analyses for Aim 2 based on all available data. Missing data will not be imputed for primary outcomes. Given the exploratory nature of the biologic outcomes and small sample size, missing values will also not be imputed. Multiple imputation will be used for missing covariates deemed necessary to adjust for in statistical modeling. Patterns of missingness will be examined as needed.

Power: Using EPDS as the continuous outcome variable compared between independent control and experimental subjects with a 1:1 allocation ratio, standard deviation of 4.89 in the control group, and true difference in mean EPDS scores of 4.00, we will need 25 subjects per group using an independent t-test to reject the null hypothesis that the population means of the groups are equal with power of 0.80 and Type 1 error probability of 0.05. To account for 20% loss to follow up, stratification, and block randomization in blocks of 2 and 4, we will enroll 44 per group for a total N=88 participants.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in English or Spanish
* Presenting for a prenatal visit with a viable singleton gestation (no known lethal fetal anomaly or plan for pregnancy termination) between 18 and 20 weeks 0 days
* Any history of depression or anxiety, defined as: 1) documented depression or anxiety in the medical record within the preceding 2 years; 2) baseline EPDS score >=10 at intake prenatal visit; 3) baseline EPDS anxiety subscale 3A score >=5

Exclusion Criteria:

* Known allergy to steel or rubber
* Implantable medical device
* Contraindication to physical activity such as a pre-existing cardiovascular condition or arrhythmia
* Plan to relocate and/or deliver at another institution
* Concurrent severe mental illness (diagnosis of bipolar disorder or schizophrenia)
* Known lethal fetal anomaly or nonviable pregnancy
* Baseline >30 min per week of vigorous physical activity (from Pregnancy Physical Activity Questionnaire, PPAQ)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Edinburgh Postpartum Depression Scale (EPDS) Score | Randomization around 20 weeks gestation and end of study (around 37 weeks gestation).
  The mean within person change in EPDS score between randomization and the end of the study will be compared between the 2 arms. The EPDS is a 10-question validated measure with a score range of 0-30 for depression and/or anxiety screening in pregnancy that has been translated into many languages. A score of >=10 has been shown to be consistent with depressive symptoms.

SECONDARY OUTCOMES:
Change in EPDS Anxiety Subscale Score | Randomization around 20 weeks gestation and end of study (around 37 weeks)
  The mean within person change in Edinburgh Postpartum Depression Anxiety Subscale score between randomization and the end of the study will be compared between the 2 arms. The three-question anxiety subscale on the EPDS (EPDS 3A) has a score range between 0-9, and a score >=5 has been shown to be consistent with anxiety symptoms.
Change in State-Trait Anxiety Inventory (STAI) Score | Randomization around 20 weeks gestation and end of study (around 37 weeks)
  Mean within person change in STAI score between randomization and the end of the study will be compared between the 2 arms. The STAI is 40 questions, and the score ranges from 40 to 160. A STAI score >=80 has been shown to be consistent with anxiety symptoms.
Change in leukocyte telomere length | Randomization around 20 weeks and end of study (around 37 weeks)
  Maternal leukocyte telomere length will be measured from saliva samples and analyzed via quantitative PCR. Mean within-person change in leukocyte telomere length will be compared between the two arms.
Change in hair cortisol level | Randomization around 20 weeks and end of study (around 37 weeks)
  Maternal hair cortisol level will be measured from consecutive segments of hair strands. Mean within-person change in hair cortisol level will be compared between the two arms.
Frequency of pregnancy complications | 6 weeks postpartum
  Frequency of pregnancy complications including hypertensive disorders, diabetes, fetal growth restriction, placental abruption, preterm birth, or stillbirth will be abstracted from the medical record
Frequency of neonatal complications | 6 weeks postpartum
  Frequency of neonatal complications including NICU admission, 5-minute Apgar <7, low birthweight, need for mechanical ventilation, or neonatal demise will be abstracted from the medical record
Neonatal leukocyte telomere length | Day of life 1
  Salivary

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Panelli, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No